CLINICAL TRIAL: NCT03460392
Title: Study of Human Microbiota in Healthy and Pathological Conditions
Acronym: MicroSP
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: MiscoSP
Record Dates: First submitted 2018-02-15; First posted 2018-03-09 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-02

CONDITIONS: Microbial Colonization
Keywords: Human microbiota
MeSH Terms: conditions — Communicable Diseases | interventions — Anti-Infective Agents; Probiotics; Cosmetics

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — * Stool samples;
  * bone and tissue biopsies;
  * tissues samples.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- Neurological and behavioral disorders: Subjects with neurological or behavioral disorders such as Tourette syndrome are enrolled.
  Interventions: Drug: Antibiotic therapy
- Subjects affected by bone diseases: Subjects affected by bone diseases such as infective osteomyelitis or osteoporosis are enrolled.
  Interventions: Drug: Antibiotic therapy
- Dysmetabolic and/or endocrine disorders: Patients with endocrine disorders, such as thyroid disfunctions, or with metabolic disorders, including diabetes mellitus,are enrolled.
- Subjects performing agonistic activity: Subjects performing physical activity at agonistic level are enrolled.
- Gastroenteric disorders: Subjects affected by gastric and/or enteric disorders are enrolled.
- Prolonged antibiotic therapy: Patients subjected to prolonged antibiotic therapies and undergone a variety of surgical procedures are enrolled.
  Interventions: Drug: Antibiotic therapy
- Healthy subjects: Subjects without any known ongoing disease are enrolled.

INTERVENTIONS:
Drug: Antibiotic therapy — To evaluate the effects of a specific event (i.e. surgical operation) or therapy (i.e antibiotic treatment) over time;
  Other Names: Probiotics, dietary factors, cosmetics and adjuvants
  Groups: Neurological and behavioral disorders; Prolonged antibiotic therapy; Subjects affected by bone diseases

SUMMARY:
The aim of the present study is to characterize the bacterial composition (microbiota) colonizing to the human body in different physio - pathological conditions (lifestyle, motor activity, surgical operations, probiotic and prebiotic consumption, antibiotic therapies, chemotherapeutic therapies), nervous and musculoskeletal diseases, gastrointestinal and metabolic disorders , oral and vaginal diseases, etc.). In particular, they will be investigate:

* the changes in the bacterial abundance
* the potential microbial interactions with the human host
* the microbial networks describing on the bacterial interactions within a specific composition of the human microbiota

DETAILED DESCRIPTION:
The main objective of this study is to deepen the knowledge about the bacterial communities associated to the human organism. In particular, the present study aims to evaluate how the microbiota (intestinal, cutaneous, vaginal, nasal, bronchial, breast milk, salivary, oral, etc.) is subject to quantitative and qualitative changes consequently to different events involving the human host. The project trys to highlight which microorganisms may be involved in the onset or progression of certain pathological condition, as well as to identify which bacterial genera can be more subject to variations due to specific non-pathological events.

Secondary objectives of this study are:

* To define a "healthy microbiome", that is to understand which are the main bacteria that commonly compose the human microbiome in physiological conditions, differentiating it from that present in certain pathological conditions.
* To characterize the physiological effects that bacterial changes of the human microbiota have on the host.
* To evaluate whether the use of probiotics, prebiotics, dietary and nutritional factors, cosmetics, and oral, nasal, vaginal, or pharmacological therapies of any kind can influence the microbial network of the human microbiota associated to different body districts.

ELIGIBILITY:
Inclusion Criteria:

* subjects suffering from neurological/behavioral diseases;
* subjects suffering of bone diseases;
* subjects affected of dysmetabolic / or endocrine disorders;
* subjects with physical activities at a competitive level;
* subjects affected of gastrointestinal disorders;
* subjects with prolonged antibiotic therapies and undergoing surgery

Exclusion Criteria:

* no use of probiotics in the month prior the sampling;
* no use of antibiotics in the month prior the sampling;
* no consumption of yogurt in the month prior the sampling;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: For each cohoort 15 healthy subjects will be enrolled (controls), for a total of 90 subjects.
  The study involves the recruitment of 180 subjects (90 pathological and 90 healthy and recruited
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-06-12 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Bacterial abundances calculated by mean of Operational Taxonomic Unit (OTU) count | Up to 24 weeks
  It is a measure of the bacterial amount

SECONDARY OUTCOMES:
Chao's indices estimated on the total OTU amount | Up to 24 weeks
  It is a measure of bacterial diversity
Simpson's index (D) estimated on the total OTU amount | Up to 24 weeks
  It is a measure of bacterial diversity
Shannon's index estimated on the total OTU amount | Up to 24 weeks
  It is a measure of bacterial diversity
The OTU abundances will be used to calculate an adjacency matrix based on the Spearman's correlation coefficient (rs) among different bacterial genus | up to 24 weeks
  It is a measure of strength of linear association between different bacterial genera

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Drago, Prof., Principal Investigator — IRCCS Galeazzi Orthopedic Institute, Milan, Italy
Locations (1):
- IRCCS Istituto Ortopedico Galeazzi, Milan, MI, Italy